CLINICAL TRIAL: NCT04915677
Title: Volumetric Changes at Edentulous Sites Augmented With Collagen Matrix or Connective Tissue Graft: a Randomized Clinical Trial With 6 Months Follow up
Brief Title: Edentulous Sites Augmented With Collagen Matrix or CTG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GFGTurin1
Record Dates: First submitted 2021-05-25; First posted 2021-06-07 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subepithelial Connective Tissue Graft (SCTG) (Active Comparator): Soft tissue augmentation at edentulous area with subepithelial connective tissue graft harvested from the patient's palate
  Interventions: Procedure: Soft tissue augmentation with subepithelial connective tissue graft (SCTG)
- Volume Stable Collagen Matrix (VCMX) (Experimental): Soft tissue augmentation at edentulous area with xenogenic volume stable collagen matrix
  Interventions: Procedure: Soft tissue augmentation with xenogenic volume stable collagen matrix

INTERVENTIONS:
Procedure: Soft tissue augmentation with subepithelial connective tissue graft (SCTG) — After local anesthesia a mesio-distal crestal incision will be performed reaching the alveolar bone. Split thickness dissection performed both buccal and palatal. Subepithelial connective tissue graft will be harvested and inserted beneath the mucoperiosteal flap and stretched buccally and lingually using a modified horizontal mattress suture. The flap margins at the crest will be adapted using single interrupted sutures in order to achieve a primary closure of the flap.
  Arms: Subepithelial Connective Tissue Graft (SCTG)
Procedure: Soft tissue augmentation with xenogenic volume stable collagen matrix — After local anesthesia a mesio-distal crestal incision will be performed reaching the alveolar bone. Split thickness dissection performed both buccal and palatal. Xenogenic volume stable collagen matrix will be inserted beneath the mucoperiosteal flap and stretched buccally and lingually using a modified horizontal mattress suture. The flap margins at the crest will be adapted using single interrupted sutures in order to achieve a primary closure of the flap.
  Arms: Volume Stable Collagen Matrix (VCMX)

SUMMARY:
Ridge deformities can complicate prosthetic rehabilitation, especially in situations where optimal esthetic outcomes are desired. Simpler, less invasive and predictable treatments are needed in order to obtain soft tissue augmentation at edentulous ridges. Autogenous subepithelial connective tissue graft (SCTG) has always been regarded as the treatment of choice, but heterologous volume stable collagen matrix (VCMX) is emerging as a reliable alternative. The principal aim of the present RCT will be to compare the volumetric buccal soft tissue changes at edentulous areas after augmentation procedure using VCMX or SCTG. Parameters related to periodontal health at adjacent teeth and patient reported outcomes (PROMs) will be also assessed as secondary outcomes. Proving the non- inferiority of VCMX compared to SCTG would provide the specialists and general clinicians with an easier, less invasive and better tolerated technique for soft tissue augmentation at edentulous ridges and for improving aesthetic and cleansability of the prosthetic rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Intercalated mono-edentulous area ridge defects to be rehabilitated with fixed partial bridge
* At least 18 years old
* At least 6 months from tooth extraction at the study area.

Exclusion Criteria:

* Systemic diseases which could influence the outcome of the therapy (e.g. uncontrolled diabetes mellitus);
* Smoking ≥ 10 cigarettes a day;
* Pregnant or nursing women;
* Chronic use of corticosteroids or other anti-inflammatory or immune-modulator drugs;
* Patients who need use of medications affecting bone metabolism or oral mucosa;
* Presence of a congruous FDP at the edentulous area;
* History of soft tissue augmentation surgery in the study area;
* Active periodontitis
* Uncompliant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-06-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Volumetric buccal soft tissue changes (-5 to +5 mm with positive values representing an increase in volume) | 6 months
  Mean linear change in mm from baseline to 6 months follow-up

SECONDARY OUTCOMES:
Change in Probing Pocket Depth (PD) at adjacent teeth (0-15 mm with higher values representing worse outcomes) | 6 months
  The distance between cementoenamel junction (CEJ) and the base of the pocket
Mucosal recession at adjacent sites (0-15 mm with higher values indicating worse outcomes) | 6 months
  The distance between the cementoenamel junction (CEJ) and the mucosal margin
Pain (VAS scale)(0-10 with higher values indicating worse outcomes) | 2 weeks
  Subjective pain experienced by the patient expressed in a VAS scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided